CLINICAL TRIAL: NCT03687268
Title: Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-centre, Phase III Trial to Investigate the Efficacy, Safety and Tolerability of Naloxone HCl PR Tablets in Patients With Opioid Induced Constipation
Brief Title: Naloxone HCl PR Tablets in Patients With Opioid Induced Constipation
Acronym: Naxos
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Develco Pharma Schweiz AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0217/DEV
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Naloxone 24 mg (Experimental)
  Interventions: Drug: Naloxone HCl PR tablets
- Naloxone 48 mg (Experimental)
  Interventions: Drug: Naloxone HCl PR tablets

INTERVENTIONS:
Drug: Naloxone HCl PR tablets — oral administration
  Arms: Naloxone 24 mg; Naloxone 48 mg
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
Prospective, randomised, double-blind, double-dummy, placebo-controlled, parallel-group, multi-centre, phase III trial of Naloxone HCl PR Tablets (12 mg and 24 mg) administered twice daily.

The trial will consist of four phases:

Screening phase (Week -4 to Week -3):

Confirmation phase (Week -2 to Week -1):

Double-blind treatment phase

Follow-up phase (Week 13-14):

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age with opioid induced constipation.
2. Long-term WHO step III opioid therapy for at least 3 months prior to screening for treatment of chronic non-cancer related pain.
3. Receiving a stable maintenance regimen with one long-acting oral or transdermal WHO step III opioid (except tapentadol) consisting of a total daily dose of ≥40 mg ME for a minimum of 4 weeks prior to screening, with no anticipated change in opioid dose requirement over the proposed trial period.
4. Symptoms of constipation with onset after the start of opioid medication for at least the last 4 weeks prior to screening,

Exclusion Criteria:

* 1. Hypersensitivity or intolerance to any active substance (i.e., naloxone, bisacodyl) or any of the excipients of the trial medication (e.g. patients with hereditary problems of galactose intolerance, lactase deficiency or glucose-galactose malabsorption). Hypersensitivity or intolerance to methylnaltrexone or naloxegol.

  2. History of cancer in the last 2 years except basal cell carcinoma and non-metastatic squamous cell skin cancer. Patients with any malignancy in the past are eligible in case they have been continuously disease-free for at least 2 years.

  3. Known or suspected reason for constipation other than OIC (e.g. idiopathic, neurological, endocrine, or metabolic).

  4. Known or suspected medical conditions that might be associated with diarrhoea, intermittent loose stools or constipation, such as faecal incontinence or irritable bowel syndrome (IBS). In case of documented suspicion of IBS or justified doubts of a long ago diagnosis, the Rome IV criteria must be applied).

  5. Any known or suspected gastrointestinal (GI) pathology that might increase the risk of perforation, such as chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis), acute diverticulitis or history of > 1 episode of diverticulitis, intestinal obstruction or pseudo-obstruction.

  6. Any form of acute temporary or permanent GI ostomy, such as ileostomy or colostomy.

  7. Renal impairment requiring any form of dialysis. 8. Known or suspected moderate-to-severe hepatic impairment (serum total bilirubin > 2 upper limit of normal (ULN) except in patients diagnosed with Gilbert's syndrome, International Normalised Ratio (INR) > 2 ULN (except in patients on therapeutic anti-coagulation), serum albumin < 2.8 g/dL) 9. Presence of any other significant or progressive/unstable medical condition that, in the opinion of the investigator, would compromise evaluation of the trial treatment or may jeopardise patient's safety, compliance or adherence to protocol requirements, such as significant psychiatric, cardiovascular, pulmonary, metabolic, endocrine or neurological disease.

  10. Any GI pathology or surgery or intractable vomiting likely to significantly influence drug absorption.

  11. Inability to swallow the trial medication whole (e.g. due to dysphagia). 12. Known or suspected acute or chronic alcoholism, delirium tremens, or toxic psychosis.

  13. Signs and symptoms that may be related to opioid withdrawal. 14. Use of prohibited medication or treatments as defined in the list of not allowed medication or treatments.

  15. For women: Pregnancy or breast-feeding. Women of childbearing potential unable or unwilling to undergo pregnancy tests and practice acceptable contraceptive measures. Acceptable methods for women are hormonal contraceptives, surgical intervention (e.g. bilateral tubal occlusion), intrauterine device, intrauterine hormone-releasing system, double-barrier methods and true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. For men: Men unable or unwilling to practice acceptable contraceptive measures. Acceptable methods for men are surgical intervention (e.g. vasectomy), true sexual abstinence and acceptable contraception (as described above) of the female partner.

  16. Previous enrolment in this trial or participation in any other drug investigational trial within the past 30 days (or five half-lives of IMP whichever is longer) prior to Visit 1 (except one re-screening in this trial).

  17. Previous treatment in a clinical trial with Naloxone HCl PR Tablets (except one re-screening in this trial).

  18. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.

  19. Employees of the investigator or trial centre, with direct involvement in the proposed trial or other studies under the direction of that investigator or trial centre, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of overall CSBM Responders. | 12 weeks
  Overall CSBM response defined as ≥ 3 CSBMs/week and an increase of ≥ 1 CSBM/week compared to baseline during at least 9 out of the 12 treatment weeks, including all of the last 4 weeks.

CONTACTS AND LOCATIONS:
Locations (104):
- Bulgaria (4):
  - Plovdiv, Plovdiv
  - Sevlievo, Sevlievo
  - Sofia, Sofia
  - Veliko Tarnovo, Veliko Tarnovo
- Czechia (12):
  - Choceň, Choceň
  - České Budějovice, České Budějovice
  - Hradec Králové, Hradec Králové
  - Liberec, Liberec
  - Most, Most
  - Ostrava, Ostrava
  - Plzeň, Pilsen
  - Praha 10, Prague
  - Sokolov, Sokolov
  - Uherské Hradiště, Uherské Hradiště
  - Zlín, Zlín
  - Znojmo, Znojmo
- Germany (15):
  - Bad Honnef, Bad Honnef
  - Bad Pyrmont, Bad Pyrmont
  - Berlin, Berlin
  - Bonn, Bonn
  - Böhlen, Böhlen
  - Eichstätt, Eichstätt
  - Fellbach, Fellbach
  - Göppingen, Göppingen
  - Hamburg, Hamburg
  - Jahnsdorf, Jahnsdorf
  - Kevelaer, Kevelaer
  - Marburg, Marburg
  - Münster, Münster
  - Stadtroda, Stadtroda
  - Würzburg, Würzburg
- Poland (13):
  - Bialystok, Bialystok
  - Bielsko-Biala, Bielsko-Biala
  - Bydgoszcz, Bydgoszcz
  - Gdansk, Gdansk
  - Katowice, Katowice
  - Krakow, Krakow
  - Lodz, Lodz
  - Ostrowiec Swietokrzyski, Ostrowiec Świętokrzyski
  - Rzeszow, Rzeszów
  - Tarnow, Tarnów
  - Tychy, Tychy
  - Warszawa, Warsaw
  - Wloclawek, Włocławek
- Portugal (8):
  - Amadora, Amadora
  - Aveiro, Aveiro
  - Braga, Braga
  - Covilhã, Covilha
  - Guimarães, Guimarães
  - Leiria, Leiria
  - Matosinhos, Matosinhos Municipality
  - Setúbal, Setúbal
- Serbia (9):
  - Belgrade, Belgrade
  - Sremska Kamenica, Kamenitz
  - Kragujevac, Kragujevac
  - Nis, Niš
  - Novi Sad, Novi Sad
  - Sombor, Sombor
  - Subotica, Subotica
  - Vrbas, Vrbas
  - Zrenjanin, Zrenjanin
- Slovakia (8):
  - Banská Bystrica, Banská Bystrica
  - Bojnice, Bojnice
  - Bratislava, Bratislava
  - Dolný Kubín, Dolný Kubín
  - Košice, Košice
  - Prešov, Prešov
  - Rimavská Sobota, Rimavská Sobota
  - Žilina, Žilina
- Spain (7):
  - Barcelona, Barcelona
  - Granada, Granada
  - Madrid, Madrid
  - Manises, Manises
  - Palma, Palma de Mallorca
  - Santiago de Compostela, Santiago de Compostela
  - Torrejón de Ardoz, Torrejón de Ardoz
- United Kingdom (28):
  - Aberdeen, Aberdeen
  - Addlestone, Addlestone
  - Belfast, Belfast
  - Chesterfield, Chesterfield
  - Clevedon, Clevedon
  - Cockermouth, Cockermouth
  - Corby, Corby
  - Dunfermline, Dunfermline
  - Durham, Durham
  - Fowey, Fowey
  - Guildford, Guildford
  - Kenilworth, Kenilworth
  - Leicester, Leicester
  - Macclesfield, Macclesfield
  - Margate, Margate
  - Middlesborough, Middlesbrough
  - Middlesex, Middlesex
  - Newcastle-Upon-Tyne, Newcastle upon Tyne
  - Northwood, Northwood
  - Penzance, Penzance
  - Plymouth, Plymouth
  - Romford, Romford
  - Salford, Salford
  - Sidcup, Sidcup
  - Sunderland, Sunderland
  - Thornton-Cleveleys, Thornton-Cleveleys
  - Wellingborough, Wellingborough
  - Wokingham, Wokingham

IPD SHARING:
Plan to Share IPD: No